CLINICAL TRIAL: NCT03908190
Title: Pilot Trial of Personalized Support for Progress (PSP) in a VA Women's Wellness Clinic
Brief Title: Personalized Support for Progress (PSP) in a VA Women's Wellness Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse VA Medical Center (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emily M. Johnson, Psychologist, Syracuse VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1297981
Record Dates: First submitted 2018-10-24; First posted 2019-04-09 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Psychological Stress; Life Stress; Emotional Stress
Keywords: Peer Support; Patient Navigators
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: The interviewer evaluating progress towards goals will be blinded to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (No Intervention): Participants will receive treatment as usual within the VHA Women's Wellness Clinic including any appropriate treatment or treatments for their medical and psychosocial concerns as determined by their primary care teams.
- Treatment As Usual Plus Personalized Support for Progress (Experimental): In addition to treatment as usual, women will receive the Personalized Support for Progress intervention.
  Interventions: Behavioral: Personalized Support for Progress

INTERVENTIONS:
Behavioral: Personalized Support for Progress — Participants will receive the Personalized Support for Progress Intervention from a peer support provider including sessions with the peer support provider to complete a prioritization task, develop a personalized care plan, and receive support for implementing the personalized care plan.
  Arms: Treatment As Usual Plus Personalized Support for Progress

SUMMARY:
The purpose of this study is to evaluate the Personalized Support for Progress (PSP) intervention in a Veterans Health Administration (VHA) Women's Wellness Clinic. PSP uses a peer support provider to help women identify their primary concern, develop a personalized plan to help address that concern, and provide practical and emotional support to implement the plan. The primary aim is to evaluate the feasibility, acceptability, and utility of PSP and the research protocol.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status (non-Veterans will not be enrolled in this trial)
* Enrollment in the Syracuse VA Medical Center Women's Wellness Clinic
* Report high stress within the last month (Perceived Stress Scale [PSS-10] > 18)
* Primary Care Provider approval for participation
* Ability to communicate in English including reading, writing, hearing, and speaking well enough to complete research and intervention tasks.

Exclusion Criteria:

* Any Veteran with "higher" suicide risk on the P4 or Veterans with "lower" suicide risk on the P4 and evaluated by the PI or another clinician to be clinically unstable or at risk
* Homicidality (screened via adaptation of the P4 screener and evaluated on the same criteria above)
* Homelessness (including literally homeless, imminent risk of homelessness, or fleeing/attempting to flee domestic violence per VA definitions)
* Veterans who are enrolled in or have had psychotherapy or changes to psychotropic medications in the last 12 weeks
* Veterans with impairment that would not allow them to engage in PSP including active psychosis, cognitive deficits, severe substance use requiring detoxification (documented in CPRS or reported by a PACT member)
* Veterans who are not available for outpatient PSP meetings (e.g., in a residential program)
* Veterans who have current VA or non-VA peer support engagement (an appointment within the last month and/or additional follow-up scheduled)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Any Veterans enrolled for care in the Syracuse VA Women's Wellness clinic because of biological sex or gender identity are eligible.
Enrollment: 28 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Assessment Retention Rate | 6 months
  This is an assessment of trial feasibility.
Intervention Retention Rate | 6 months
  This is an assessment of trial feasibility.
Client Satisfaction Questionnaire | 6 months
  This scale measures satisfaction and ranges from 8-24 with higher scores indicating higher satisfaction.
Goal Attainment Scaling | 6 months
  This interview assesses progress toward individualized goals on a -2 to 2 scale with higher scores indicating more progress toward goals.
Perceived Stress Scale (PSS-10) | 6 months
  This scale evaluates perceived stress and ranges from 0-40 with lower scores indicating lower levels of perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse VA Medical Center, Syracuse, New York, United States